CLINICAL TRIAL: NCT05388682
Title: Observation of Long Term Effect of Medical and PTPA Treatment on Patients With Takayasu Arteritis Complicated With Pulmonary Artery Involvement
Brief Title: Treatment of Patients With Takayasu Arteritis Complicated With Pulmonary Artery Involvement
Status: Recruiting | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: TAPAI
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-01

CONDITIONS: Takayasu Arteritis With Pulmonary Artery Involvement; Percutaneous Transluminal Pulmonary Angioplasty; PAH Targeted Medication
Keywords: Percutaneous transluminal pulmonary angioplasty, Takayasu Arteritis with Pulmonary Artery Involvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous transluminal pulmonary angioplasty — Percutaneous transluminal pulmonary angioplasty

SUMMARY:
1. Evaluate the effect of medical treatment and percutaneous transluminal pulmonary angioplasty on takayasu arteritis with pulmonary artery involvement
2. evaluate the efficacy of FAPI in predicting the activity and treatment efficacy of takayasu arteritis with pulmonary artery involvement

DETAILED DESCRIPTION:
At baseline, FAPI and FDG are performed to evaluate the activity of takayasu arteritis with pulmonary artery involvement. FAPI is also used to predict the treatment efficacy and prognosis of takayasu arteritis with pulmonary artery involvement.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Takayasu arteries with pulmonary arteries involvement

Exclusion Criteria:

* Patients had pulmonary artery stenosis arising from CTEPH, fibrosing mediastinitis and congenital pulmonary artery stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with Takayasu arteries with pulmonary arteries involvement received either medical or percutaneous transluminal pulmonary angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01-19 (Actual); Primary Completion 2042-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
all cause death | 2014/1/1-2042/12/31
  all cause death
mean pulmonary arterial pressure change | 2014/1/1-2042/12/31
  change of mean pulmonary arterial pressure after treatment
pulmonary vascular resistance change | 2014/1/1-2042/12/31
  chagne of pulmonary vascular resistance after treatment
6MWD change | 2014/1/1-2042/12/31
  change of six minute walk distance after treatment
peak VO2 change | 2014/1/1-2042/12/31
  change of peak oxygen consumption after treatment
NT-proBNP change | 2014/1/1-2042/12/31
  change of NT-proBNP after treatment
RV/LV change | 2014/1/1-2042/12/31
  change of right ventricular end-diastolic diameter versus laboratory left ventricular end-diastolic diameterafter treatment
CI change | 2014/1/1-2042/12/31
  change of cardiac index after treatment

CONTACTS AND LOCATIONS:
Overall Officials: zhihong Liu, doctor, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No